CLINICAL TRIAL: NCT01759524
Title: To Compare lidocaine2%/Clonidine in Combination With Bupivacaine 0.5 % Alone in Equal Volumes for Combined Sciatic-saphenous Nerve Block in Terms of Selectivity of Blockade
Brief Title: To Compare lidocaine2%/Clonidine in Combination, With Bupivacaine 0.5 % Alone in Equal Volumes for Combined Sciatic-saphenous Nerve Block in Terms of Selectivity of Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, DR. Jassim Rauf, Clinical Research/ Peripheral Nerve Blocks Fellow., Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JR-786-GS
Record Dates: First submitted 2012-12-27; First posted 2013-01-03 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Bimalleolar Fractures of the Ankle.; Sciatic Nerve Block.; Saphenous Nerve Block.; Post Operative Analgesia Duration.
Keywords: local anaesthesia; analgesia; bupivacaine; lidocaine; clonidine; sciatic nerve; saphenous nerve
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Lidocaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group L (Experimental): 40 mls of 2% lidocaine + 1.5 mcg/kg will be drawn up by an attending anaesthetist to blind the operator. Patients in this group will receive an ultra sound guided sciatic nerve block , 3 cm proximal to the nerve bifurcation, with 25 mls of the above mentioned solution and an ultra sound guided saphenous nerve block in the midthigh just lateral to the profunda femoris artery with 15 mls of the above mentioned solution.
  Interventions: Drug: Lidocaine
- Group B (Active Comparator): 40 mls of 0.5% bupivacaine will be drawn up by an attending anaesthetist to blind the operator. Patients in this group will receive an ultra sound guided sciatic nerve block , 3 cm proximal to the nerve bifurcation, with 25 mls of the above mentioned solution and an ultra sound guided saphenous nerve block in the midthigh just lateral to the profunda femoris artery with 15 mls of the above mentioned solution.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine
  Other Names: 0.5% bupivacaine, marcaine.
  Arms: Group B
Drug: Lidocaine
  Other Names: 2% lidocaine + 1.5 mcg/kg clonidine
  Arms: Group L

SUMMARY:
Clonidine as an adjuvant to local anaesthetics prolongs the postoperative analgesia. It is predominantly an alpha 2 agonist, but does have some alpha 1 activity. Clonidine alone produces analgesia. When administered centrally its effects are predominantly due to its alpha 2 activity. When administered peripherally it prolongs the analgesia through its vasoconstrictor effects and by reducing the clearance of local anaesthetic. Another possibility is that it prolongs analgesia of peripheral nerve blocks due to a hyperpolarisation current .Clonidine has been used successfully both for upper and lower limb blocks. Studies of clonidine for lower limb blocks have produced equivocal results . A major concern with the lower limb blocks is the risk of falls associated with prolonged motor blockade during early mobilisation. Clonidine has been shown to intensify and prolong the motor blockade produced by long acting local anaesthetics. Lidocaine when used in combination with clonidine can increase the duration of analgesia to 8-18 hrs. Greater doses of clonidine are associated with longer analgesia but with more side effects. Clonidine in a dose of 90 mcg administered with local anaesthetics can produce analgesia for up to 10 hrs with minimal side effects. The aim of this study is to compare lidocaine 2% + clonidine 1.5mcg/kg with bupivacaine alone in terms of block selectivity for combined sciatic -saphenous nerve block in patients under going semi elective foot/ankle procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients scheduled to undergo semi elective ankle/foot surgery with regional anaesthesia will be recruited.

Exclusion Criteria:

* patient refusal,
* allergy to local anaesthetics,
* coagulopathy,
* malignancy or infection at the block performance site,
* significant peripheral neuropathy or neurologic disorder of the lower extremity or any other contraindication to sciatic and saphenous nerve block,
* pregnancy,
* history of alcohol or drug dependency/abuse (defined as >40 IU/week),
* a history of significant cognitive or psychiatric disorder that may affect patient assessment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative sensory and motor block. | 36 hours.
  Postoperative analgesia/duration of block will be assessed at 4,6 8, 10,12,16 hrs or until complete recovery of sensation to cold spray upto 36 hours.

SECONDARY OUTCOMES:
Onset time of block. | every 5 minutes upto 40 minutes
  After completion of the two blocks the effect will be assessed every 5 minutes for onset time defined as the time from withdrawal of needle (t0) to complete loss of sensation in the sensory dermatomes of both sciatic and saphenous nerve.
  The sensory level will be assessed on toes and forefoot due to post operative cast restricted access to full tibial and peroneal nerve dermatomes.
  Motor block assessment will carried out using bromage and modified bromage scale for tibial and peroneal nerve

CONTACTS AND LOCATIONS:
Overall Officials: George Shorten, FCARCSI PhD, Study Chair — Cork University Hospital, Cork, Ireland.
Locations (1):
- Cork University Hospital, Cork, Ireland